CLINICAL TRIAL: NCT01559675
Title: Randomized Controlled Trial Comparing Low Dose and High Dose Steroids in Patients Undergoing Colorectal Surgery
Brief Title: Trial Comparing Low Dose and High Dose Steroids in Patients Undergoing Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Fleshner MD, Colon & Rectal Surgeon, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSMCSteroidStudy
Record Dates: First submitted 2012-03-16; First posted 2012-03-21 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Orthostatic Hypotension; Hemodynamic Instability; Fever; Hypothermia
Keywords: Corticosteroids; perioperative; colorectal surgery
MeSH Terms: conditions — Hypotension, Orthostatic; Fever; Hypothermia | interventions — Hydrocortisone; Methylprednisolone Hemisuccinate; Adrenal Cortex Hormones; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrocortisone High Dose (Active Comparator): Intervention: Patients receive Hydrocortisone 100 mg at surgical incision followed by 100mg IV every 8 hours for the first 24 hours, followed by 75 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 12 hours, followed by Prednisone 20 mg orally when oral diet is resumed
  Interventions: Drug: Hydrocortisone High Dose
- Hydrocortisone Low Dose (Experimental): Intervention: 1/3 Intravenous equivalent dose (IVED) at surgical incision, followed by 1/3 IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD) 1, followed by 1/6 IVED every 8 hours on POD 2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
  Interventions: Drug: Hydrocortisone Low Dose

INTERVENTIONS:
Drug: Hydrocortisone High Dose — Patients receive Hydrocortisone 100 mg at surgical incision followed by 100mg IV every 8 hours for the first 24 hours, followed by 75 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 12 hours, followed by Prednisone 20 mg orally when oral diet is resumed
  Other Names: Solumedrol; Corticosteroid; Steroid
  Arms: Hydrocortisone High Dose
Drug: Hydrocortisone Low Dose — 1/3 IV equivalent dose (IVED) (hydrocortisone equivalent of the patient's preoperative steroid dose) at surgical incision, followed by 1/3 IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD 2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
  Other Names: Solumedrol; Corticosteroid; Steroid
  Arms: Hydrocortisone Low Dose

SUMMARY:
The purpose of this study is to evaluate the effect of low dose versus high dose steroids vital signs of patients currently on steroids or recently treated with steroids undergoing major colorectal surgery. The investigators hypothesize that there will be no statistically significant difference in orthostatic hypotension (blood pressure measured on lying, sitting, and standing), blood pressure, temperature or heart rate in the standard and low dose groups.

DETAILED DESCRIPTION:
Our primary aim is to study the perioperative hemodynamic profile of patients on chronic steroids undergoing colon and rectal surgery. We will do this by measuring heart rate, temperature and blood pressure in the operating room and during their postoperative hospitalization. Patients will be identified in their preoperative visit. They will be randomized to high dose and low dose steroid study groups. The standard dose steroid patients will receive hydrocortisone 100 mg IV preoperatively and 100 mg IV every 8 hrs with standard taper. The low dose steroid study group will receive the IV equivalent of their preoperative steroid dose in the postoperative period. The patients blood pressure, temperature and heart rate will be monitored in the operating room and the ward postoperatively. Outcomes will be compared between the two groups. We hypothesize that there will be no statistically significant difference in blood pressure, temperature or heart rate in the high dose and low dose groups.

The secondary aim of this study will be monitoring of any differences in surgical outcomes, including postoperative length of stay, between the two patient groups.

ELIGIBILITY:
Inclusion Criteria:

* History of ulcerative colitis, inflammatory bowel disease unclassified, indeterminate colitis, or Crohn's disease;
* Major colorectal surgery, defined as surgery requiring an abdominal incision. Both open and laparoscopic procedures are eligible. Urgent and elective procedures are eligible;
* Corticosteroid therapy within 12 months of surgery;
* Able and willing to comply with all protocol procedures for the planned duration of the study
* Able and willing to understand, sign and date an informed consent document, and authorize access to protected health information.

Exclusion Criteria:

* Patients with hypotension (systolic < 90 mm Hg or diastolic < 50 mm Hg) in the preoperative area
* Patients having emergency surgery
* Children < 18 or adults > 75 years of age
* Pregnant patients
* Patients who have suffered prior hemodynamic complications of steroid withdrawal
* Other major physical or major psychiatric illness, including alcohol or substance addiction, within the last 6 months that in the opinion of the investigator would affect the patient's ability to complete the trial.
* Any condition or situation that, in the opinion of the investigator, would prevent proper evaluation of the safety or efficacy of the different steroid doses according to the study protocol
* Patients on steroids without inflammatory bowel disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Fleshner, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Zaghiyan K, Melmed GY, Berel D, Ovsepyan G, Murrell Z, Fleshner P. A prospective, randomized, noninferiority trial of steroid dosing after major colorectal surgery. Ann Surg. 2014 Jan;259(1):32-7. doi: 10.1097/SLA.0b013e318297adca. PMID 23774314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2010 and March 2012, 121 patients with Inflammatory bowel disease (IBD) between the ages of 18 to 75 years taking corticosteroids, or previously treated with steroids within the previous 1 year, undergoing major colorectal surgery by a single surgeon at a single institution were recruited for this study
Pre-assignment Details: Of 258 patients assessed for eligibility, 137did not meet inclusion criteria. 9 patients refused to participate. 121 were then randomized to one of 2 study arms
Groups:
- High Dose Steroid: Patients receive Hydrocortisone 100 mg at surgical incision followed by 100mg IV every 8 hours for the first 24 hours, followed by 75 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 12 hours, followed by Prednisone 20 mg orally when oral diet is resumed
  Hydrocortisone: Patients receive Hydrocortisone 100 mg at surgical incision followed by 100mg IV every 8 hours for the first 24 hours, followed by 75 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 8 hours for 24 hours, followed by 50 mg IV every 12 hours, followed by Prednisone 20 mg orally when oral diet is resumed
- Low Dose Steroid: 1/3 Intravenous equivalent dose (IVED) at surgical incision, followed by 1/3 IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD 2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
  Hydrocortisone: 1/3 IV equivalent dose (IVED) (hydrocortisone equivalent of the patient's preoperative steroid dose) at surgical incision, followed by 1/3IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
Period: Overall Study
Arm/Group | High Dose Steroid | Low Dose Steroid
Started | 58 | 63
Completed | 43 | 49
Not Completed | 15 | 14
Not completed — Protocol Violation | 1 | 2
Not completed — 2nd operation on same patient excluded | 14 | 12

BASELINE CHARACTERISTICS:
Population: We assumed that patients treated with HDS would have no postural hypotension on POD1 95% of the time. The noninferiority margin was 10%. We calculated that a sample size of 118 patients (59 patients per study arm) was needed to establish clinical equivalency with a 1-sided α level of 0.05 and 80% power.
Groups:
- Low Dose Steroid: 1/3 Intravenous equivalent dose (IVED) at surgical incision, followed by 1/3 IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
  Hydrocortisone: 1/3 IV equivalent dose (IVED) (hydrocortisone equivalent of the patient's preoperative steroid dose) at surgical incision, followed by 1/3 IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD 2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
- Total: Total of all reporting groups
Arm/Group | High Dose Steroid | Low Dose Steroid | Total
Number analyzed (Participants) | 43 | 49 | 92
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [24 to 50] | 41 [29 to 50] | 40 [24 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 22 | 27 | 49

OUTCOME MEASURES:

1. Primary Outcome: Orthostatic Hypotension
Time Frame: Postoperative Day 1
Measure: Number; unit: participants
Groups:
- Low Dose Steroid: 1/3 Intravenous equivalent dose (IVED) at surgical incision, followed by 1/3IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
  Hydrocortisone: 1/3 IV equivalent dose (IVED) (hydrocortisone equivalent of the patient's preoperative steroid dose) at surgical incision, followed by 1/3IVED for 24 hours, Patients subsequently treated with 1/4 IVED every 8 hours starting Postoperative day (POD 1), followed by 1/6 IVED every 8 hours on POD2 and every 12 hours starting POD 3. On POD 4 or when the patient was tolerating a regular diet, oral prednisone equal to the most recent IV hydrocortisone dose resumed
Arm/Group | High Dose Steroid | Low Dose Steroid
Number analyzed (Participants) | 43 | 49
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: adverse events were collected for the 30-day postoperative period.
Description: adverse events were identified through patient chart review, reporting by investigators, and at the time of patient follow up for postoperative followup and phone call at 30 days
Arm/Group | High Dose Steroid | Low Dose Steroid
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/49
Other Adverse Events (participants affected / at risk) | 11/43 | 12/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Steroid (N=43) | Low Dose Steroid (N=49)
Minor surgical complication (Gastrointestinal disorders) | 2 | 3
Major surgical complication (Gastrointestinal disorders) | 6 | 7
Major Medical complication (Cardiac disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No